CLINICAL TRIAL: NCT02392689
Title: Improve Management of Heart Failure With Procalcitonin - Biomarkers in Cardiology 18
Brief Title: Improve Management of Heart Failure With Procalcitonin
Acronym: IMPACT-EU
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: At 75% patient completion overall mortality was much lower than expected and without significant difference at day 90. No chance to reach the primary endpoint.
Sponsor: Brahms AG (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: IMPACT-EU
Record Dates: First submitted 2015-03-09; First posted 2015-03-19 (Estimated); Last update posted 2018-07-23 (Actual); Status verified 2018-07

CONDITIONS: Heart Failure; Infection
Keywords: procalcitonin; biomarker; antibiotic therapy; emergency department; cardiology; in vitro diagnostics
MeSH Terms: conditions — Heart Failure; Infections; Emergencies | interventions — Procalcitonin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- PCT-guided (Experimental): Blood samples are taken on day 0 and day 1 of the study. Procalcitonin (PCT) is measured and used support the decision on antibiotic therapy.
  PCT levels above 0.2 ng/ml: antibiotic therapy is recommended PCT levels equal/below 0.2 ng/ml: antibiotic therapy is not recommended
  Interventions: Other: Procalcitonin
- Standard of Care (No Intervention): Blood samples are taken on day 0 and day 1 and stored for later analysis. The investigator treats the patients according to standard of care.

INTERVENTIONS:
Other: Procalcitonin — Procalcitonin guided antibiotic therapy
  Arms: PCT-guided

SUMMARY:
Patients presenting to the Emergency Department with shortness of breath and (suspected) heart failure will be screened and randomized to either a standard of care or a procalcitonin-guided arm.

Procalcitonin-guided arm: a procalcitonin level (cutoff 0.2 ng/ml) will be used to support decision on antibiotic therapy initiation.

Standard of care arm: the decision on antibiotic therapy will be based on the physicians intent to treat.

The patients will be followed up 30 and 90 days after randomization to evaluate the survival status, re-hospitalizations and further antibiotic therapies.

ELIGIBILITY:
Inclusion Criteria:

1. Patients who present to the emergency department (ED) with leading symptom dyspnea
2. Suspected or known heart failure
3. midregional pro atrial natriuretic peptide (MR-proANP)>300 pmol/L, brain natriuretic peptid (BNP) >350 ng/ml or N-terminal of the prohormone brain natriuretic peptide (NT-proBNP)>1800 ng/l
4. Patient has given written Informed Consent within study timelines to allow antibiotic therapy within 8 hours
5. Adult patients (i.e. >18 years of age)
6. Hospitalization for at least 1 overnight stay planned

Exclusion Criteria:

1. Patient participates in any other interventional clinical trial
2. Trauma related shortness of breath
3. Patient diagnosed with lung or thyroid cancer
4. Known terminal disease with life expectancy of less than 6 months, e.g. advanced metastasized cancer disease
5. Organ transplant requiring immunosuppression
6. Abdominal, vascular or thorax surgery within the last 30 days
7. End stage/advanced heart failure - defined by planned heart transplantation, or cardiogenic shock
8. Female patients who have given birth within 3 months before study enrolment
9. Current use of antibiotics or requirement of immediate antibiotic therapy before randomization and measurement of Procalcitonin
10. End stage renal failure requiring dialysis
11. Patient is not willing, or it is not possible or advisable for the patient, to follow the study schedule, including antibiotic therapy and 90 days follow up
12. Patient has already participated in the clinical trial previously
13. Pregnant or lactating women
14. Patients who are institutionalized by official or judicial order
15. Dependants of the sponsor, the contract research organization (CRO), the study site or the investigator

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 759 (Actual)
Dates: Start 2015-03 (Actual); Primary Completion 2018-04-05 (Actual); Study Completion 2018-04-14 (Actual)

PRIMARY OUTCOMES:
all cause mortality | 90 days

SECONDARY OUTCOMES:
all cause mortality | 30 days
all-cause hospital readmission | 30 days
Number of patients with diagnosis of pneumonia during index hospitalization | participants will be followed for the duration of hospital stay, an expected average of 1 week

CONTACTS AND LOCATIONS:
Overall Officials: Alan Maisel, MD, Principal Investigator — University of California-San Diego/VA San Diego Healthcare System; Martin Möckel, MD, Principal Investigator — university hospital Charitè Berlin
Locations (15):
- Denmark (3):
  - Aalborg Sygehus, Aalborg
  - Herlev Hospital, Herlev
  - Odense University Hospital, Odense
- Germany (9):
  - Kerckhoff-Klinik, Bad Nauheim
  - Charite Universitätsmedizin Berlin - CCM, Berlin
  - Charite Universitätmedizin Berlin - CVK, Berlin
  - Universitätsklinikum Frankfurt, Frankfurt am Main
  - Klinikum Frankfurt Höchst GmbH, Frankfurt am Main
  - Universitätsmedizin Göttingen, Göttingen
  - Medizinische Universitätsklinik Heidelberg - Medizinische Klinik III, Heidelberg
  - Universitäres Herzzentrum Lübeck, Lübeck
  - Klinikum Nürnberg Nord, Nuremberg
- Netherlands (2):
  - University Medical Center Groningen, Groningen
  - Maastricht UMC+, Maastricht
- Hospital Clinico San Carlos, Madrid, Spain